CLINICAL TRIAL: NCT01868035
Title: Phase II Multicenter Study of Iodine-131 Anti-B1 Antibody Consolidation For Patients With Diffuse Large B-Cell Non-Hodgkin's Lymphoma Following First-line CHOP
Brief Title: Iodine-131 Anti-B1 Antibody Consolidation for Patients With Non-Hodgkin's Lymphoma Following First-line CHOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 393229/007
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Results first posted 2013-09-12 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: radioimmunotherapy; Iodine 131 Tositumomab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): tositumomab and iodine I-131 tositumomab
  Interventions: Drug: tositumomab and iodine I-131 tositumomab

INTERVENTIONS:
Drug: tositumomab and iodine I-131 tositumomab — Subjects received the following treatments of TST/I-131 TST by intravenous (IV) infusion:
  Dosimetric Dose: 450 mg of TST infused over 1 hour immediately followed by 35 mg of TST labeled with 5 milliCuries (mCi) of I 131 infused over 30 minutes.
  Therapeutic Dose: 7 to 14 days after the dosimetric dose, 450 mg of TST infused over 60 minutes, immediately followed by 35 mg of TST labeled with the subject-specific mCi activity of I 131 needed to deliver a total body dose of 75 centiGrays (cGy), infused over 30 minutes for subjects with a platelet count of 150,000/mm3. Subjects with platelet counts of 100,000 to 149,999/mm3 received 65 cGy, and obese subjects were dosed based upon 137% of their calculated lean body mass.
  Other Names: Bexxar

SUMMARY:
This is a multicenter study for the long-term follow-up of surviving patients who are expected to complete or who have completed at least two years of follow-up after treatment with Iodine I 131 Tositumomab (BEXXAR) on studies CP-97-011, CP-98-025, CP-99-032, or CP-99-036. All patients will be assessed for survival and disease status, including subsequent therapy for Diffuse Large B-cell Non-Hodgkin's Lymphoma (NHL), and for long-term safety. Additionally laboratory evaluations consisting of a thyroid stimulating hormone (TSH) level and a complete blood cell (CBC) count with a differential and platelet count will be obtained annually. Additionally, patients who remain in long-term response following Iodine I 131 Tositumomab treatment will be followed for response and progression.

DETAILED DESCRIPTION:
This is a phase II, open-label, multicenter study of Iodine-131 Anti-B1 Antibody consolidation for 20 patients with diffuse large B-cell non-Hodgkin's lymphoma (NHL) achieving a partial response (PR), an unconfirmed complete response (CRu), or complete response (CR) following 6-8 cycles of first-line cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) chemotherapy. Although the majority of patients entered in previous Iodine-131 Anti-B1 Antibody studies had low-grade or transformed low-grade NHL, 15 patients with de novo intermediate-grade NHL have been treated. Patients will undergo two dosing phases of Iodine-131 Anti-B1 Antibody.

In the first phase, termed the "dosimetric dose," patients will receive an infusion of unlabeled Anti-B1 Antibody (450 mg) over 60 minutes followed by a 30-minute infusion (including a 10-minute flush) of Anti-B1 Antibody (35 mg) that contains 5 mCi of Iodine-131. Whole body gamma camera scans will be obtained on Day 0; Day 2, 3, or 4; and Day 6 or 7 following the dosimetric dose. Using the dosimetric data from the three imaging time points, a patient-specific dose of Iodine-131 will be calculated to deliver the desired total body dose of radiotherapy. In the second phase, termed the "therapeutic dose," patients will receive a 60-minute infusion of unlabeled Anti-B1 Antibody (450 mg) followed by a 30-minute infusion (including a 10-minute flush) of 35 mg Anti-B1 Antibody labeled with a patient-specific dose of Iodine-131 calculated to deliver a 75 cGy total body radiation dose . Patients who have platelet counts of 100,000-149,999 cells/mm3 will receive 65 cGy and patients who are obese will be dosed based upon 137% of their lean body mass. Patients will be treated with saturated solution potassium iodide (SSKI), Lugol's solution, or potassium iodide tablets starting at least 24 hours prior to the first infusion of the Iodine-131 Anti-B1 Antibody (i.e., dosimetric dose) and continuing for 14 days following the last infusion of Iodine-131 Anti-B1 Antibody (i.e., therapeutic dose).

The primary endpoint of this study is to determine the incidence of Grade IV hematologic toxicity following Iodine-131 Anti-B1 Antibody consolidation for patients with diffuse large B-cell NHL who achieved a response (PR, CRu, CR) following first-line CHOP chemotherapy. The secondary efficacy endpoints are to determine the complete response rate, duration of response, duration of complete response, progression-free survival, and time to treatment failure. The pharmacokinetic endpoint is to determine the total body residence time following the dosimetric dose. The secondary safety endpoints are to determine the incidence of adverse experiences, hematologic toxicity (e.g., nadir, time to nadir, and time to recovery), use of supportive care, percent of patients converting to human anti-murine antibody (HAMA) positivity, and survival.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects age 18 to 80 years, inclusive, with any International Prognostic Index score; treated with 6 or more cycles of first-line CHOP chemotherapy and achieved a PR, CRu, or CR
* de novo diffuse large B-cell NHL according to the REAL classification; Ann Arbor stage III, stage IV, or bulky stage II disease (any mass ≥10 cm in diameter)
* less than an average of 25% of the intratrabecular marrow space involved by NHL in bilateral bone marrow biopsy specimens or <10% involvement with NHL from unilateral bone marrow biopsy; tumor tissue expressing the CD20 antigen
* ≥60% performance status on the Karnofsky Performance Scale and an anticipated survival of at least 3 months
* absolute neutrophil count (ANC) ≥1500 cells/mm3 and platelet count ≥100,000/mm3
* adequate renal function (serum creatinine <1.5 × upper limit of normal [ULN]) and hepatic function (total bilirubin ≤2.0 × ULN and aspartate aminotransferase <5 × ULN)

Exclusion Criteria:

* prior radiation, prior biological therapy, or prior chemotherapy other than first-line CHOP
* active bilateral obstructive hydronephrosis
* New York Heart Association class III or IV heart disease or other serious illness
* prior malignancy other than lymphoma (except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which they had been disease-free for >5 years)
* human immunodeficiency virus infection
* HAMA positive
* brain or leptomeningeal metastases at any time since diagnosis
* active infection requiring intravenous anti-infectives
* pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Leonard JP, Gregory SA, Smith H, Horner TJ, Williams VC, Giampietro P, Lin TS. CHOP Chemotherapy Followed by Tositumomab and Iodine-131 Tositumomab for Previously Untreated Diffuse Large B-cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2016 Apr;16(4):191-6. doi: 10.1016/j.clml.2015.12.011. Epub 2016 Jan 4. PMID 26832194
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 393229/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 393229/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 393229/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 393229/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 393229/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 393229/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 393229/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were treated with 6 to 8 cycles of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) therapy, and were required to have a response (complete response [CR], complete response unconfirmed [CRu], partial response [PR]) to be eligible for Tositumomab and iodine I 131 tositumomab (TST/I 131 TST) therapy.
Groups:
- TST/Iodine I-131 TST: Participants received an infusion of 450 milligrams (mg) of unlabeled Anti-B1 antibody of Tositumomab (TST) over the course of 60 minutes, followed by a 30 minute infusion (including a 10 minute flush) of 35 mg Anti-B1 antibody of TST labelled with 5 miillicuries (5 mCi) of Iodine-131.
Period: Overall Study
Arm/Group | TST/Iodine I-131 TST
Started | 15
Completed | 8 (These participants completed 10 years of follow-up.)
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 2
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (13.9)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13
  Hispanic | 1
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Grade 4 Hematology Toxicities Following Iodine-131 Anti-B1 Antibody
Description: Hematology parameter grades were summarized according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 2.0. Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening or disabling; Grade 5, death. Data are presented for those participants who experienced Grade 4 toxicities. Grade 4 hematological toxicities included absolute neutrophil count (ANC) (calculated) <1000 cells/millimeters cubed (mm^3), white blood cells (WBC) <2000 cells/mm^3, platelets <50000 cells/mm^3, and hemoglobin < 8.0 grams/deciliter.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: Intent-to-treat (ITT) Population: all participants who received study drug
Measure: Number; unit: participants
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
participants
  ANC (calculated) | 1
  WBC count | 1
  Platelet count | 1
  Hemoglobin | 1

2. Secondary Outcome: Number of Participants (Par.) With Confirmed (Con.) Complete Response (CR) Confirmed, Confirmed Complete Response Unconfirmed (CRu), Confirmed Partial Response (PR), Relapse Disease (RD), and Progressive Disease (PD)
Description: CR is defined as the complete disappearance of all detectable clinical/radiographic evidence of disease, the disappearance of all disease-related symptoms if present before therapy, and normalization of biochemical abnormalities definitely assignable to non Hodgkin's lymphoma (NHL). PR is defined as a >=50% decrease in the sum of perpendicular diameters (SPPD) of splenic and hepatic nodules determined at Baseline. SD is defined as less than a PR, but not PD, which is defined as a >=50% increase from nadir in SPPD of splenic and hepatic nodules or the appearance of any new lesion during or at the end of therapy that was >1.5 centimeters (cm) by radiographic evaluation or >1.0 cm by physical examination. RD is defined as the appearance of any new lesion or an increase of >= 50% in the size of nodules. Confirmed response requires that the same or better response be confirmed by two consecutive post-therapy response evaluations at least 4 weeks apart.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population. A con. CR+CRu requires that the best response be con. by the same response or better >=4 weeks apart. The individual rows for con. CR, CRu, and PR represent par. with the best response con. by the same exact response. One par. in the CR+CRu category is not counted in the con. CR category because the CR was not con. by another CR.
Measure: Number; unit: participants
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
participants
  CR | 12
  CRu | 0
  CR + CRu | 13
  PR | 1
  SD | 0
  PD | 0

3. Secondary Outcome: Duration of Response and Duration of Confirmed Complete Response
Description: Duration of response for all participants with confirmed PR, confirmed CRu, or confirmed CR is defined as the time from the first documented response to the first documented progression. CR is defined as the complete disappearance of all detectable clinical/radiographic evidence of disease, the disappearance of all disease-related symptoms if present before therapy, and the normalization of biochemical abnormalities definitely assignable to NHL. PR is defined as a >=50% decrease in the sum of the perpendicular diameters (SPPD) of splenic and hepatic nodules determined at Baseline. PD is defined as a >=50% increase from nadir in SPPD of splenic and hepatic nodules or the appearance of any new lesion during or at the end of therapy that was >1.5 centimeters (cm) by radiographic evaluation or >1.0 cm by physical examination. Confirmed response requires that the same or better response be confirmed by two consecutive post-therapy response evaluations at least 4 weeks apart.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population. Only those participants with a confirmed response were analyzed. Duration measures were calculated using Kaplan-Meier techniques.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 14
months
  All confirmed responders, n=14 | 58.4 [12.0 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval due to the low number of events.
  Confirmed complete responders, n=12 | 58.4 [20.9 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval due to the low number of events.

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the start of treatment to the first documented progression or death. Duration measures were calculated using Kaplan-Meier techniques. Disease progression was based on radiographic or photographic evidence, and assessments were made by the investigator. PD is defined as a >=50% increase from nadir in SPPD of splenic and hepatic nodules or the appearance of any new lesion during or at the end of therapy that was >1.5 centimeters (cm) by radiographic evaluation or >1.0 cm by physical examination.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
months | 63.0 [16.1 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval due to the low number of events.

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as the time from the start of treatment to the first occurrence of treatment withdrawal, decision to seek additional therapy, study removal, disease progression, or death. Duration measures were calculated using Kaplan-Meier techniques. Disease progression was based on radiographic or photographic evidence, and assessments were made by the investigator. PD is defined as a >=50% increase from nadir in SPPD of splenic and hepatic nodules or the appearance of any new lesion during or at the end of therapy that was >1.5 centimeters (cm) by radiographic evaluation or >1.0 cm by physical examination.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
months | 63.0 [16.1 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval due to the low number of events.

6. Secondary Outcome: Total Body Residence Time (TBRT)
Description: TBRT is the time at which the activity of infusion is 37% of that at time zero. Whole body images from anterior and posterior gamma camera scans were collected to assess dosimetry. The assessment of organ dosimetry required gamma camera scans from at least 4 time points. Nuclear medicine reviewers conducted a visual examination of the gamma camera scans and calculated the TBRTs. Residence time is calculated from the rate of total body clearance of iodine I-131 radioactivity during the dosimetric dose. Residence time is a measure of how long the drug resides in the body.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
hours | 105.5 (11.55)

7. Secondary Outcome: Number of Participants With an Adverse Experience, Including Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and does not necessarily have to have a casual relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or significant worsening of a pre-existing sign or symptom, or disease temporally associated with the use of a medicinal product. An SAE is defined as any experience occurring at any dose that results in the following outcomes: death, a life-threatening adverse experience, in-patient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. See the SAE/AE module for a complete list of SAEs/AEs.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
participants
  Any AE | 14
  Any SAE | 3

8. Secondary Outcome: Time to Recovery From the Indicated Hematology Toxicities
Description: Hematology toxicities included ANC (calculated), WBC count, platelet count, and hemoglobin. Time to recovery to Baseline grade for participants with Grade 0 toxicity at Baseline was defined as the time from the date of the last administration of study drug to the first post-nadir date with Grade 0 toxicity, with no other Grade 1-4 toxicities recorded during the next week. For participants with a Grade 1-4 toxicity at Baseline, time to recovery was defined as the time from the last administration of study drug to the first post-nadir date with a Baseline grade or better, with no other higher grade toxicities recorded during the next week. For participants with a nadir grade less than or equal to the Baseline grade, the time to recovery to the Baseline grade equaled the time to nadir.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
days
  ANC (calculated) | 78.5 [57.0 to 90.0]
  Hemoglobin | 69.0 [41.0 to 167.0]
  Platelet count | 51.0 [43.0 to 70.0]
  WBC count | 77.0 [71.0 to 91.0]

9. Secondary Outcome: Nadir for the Indicated Hematology Toxicities
Description: Hematology toxicities included ANC (calculated), hemoglobin, platelet count, WBC count. Nadir is defined as lowest counts that the cells reach after chemotherapy.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: 10^3 cells/millimeters cubed (mm^3)
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
10^3 cells/millimeters cubed (mm^3)
  Nadir, Baseline, ANC | 1.1 (0.47)
  Nadir, Baseline, Hemoglobin | 10.5 (2.37)
  Nadir, Baseline, platelet count | 89.9 (45.85)
  Nadir, Baseline, WBC count | 2.2 (0.70)

10. Secondary Outcome: Time to Nadir for the Indicated Hematology Toxicities
Description: Hematology toxicities included ANC (calculated), WBC count, platelet count, and hemoglobin. Nadir is defined as the lowest counts (for ANC, WBC, and platelet counts)/concentration (for hemoglobin) that the cells reach after chemotherapy. Time to nadir is defined as the time from Baseline to the lowest value recorded up to 120 days following the therapeutic dose.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
days
  Time to nadir, ANC | 55.0 (16.52)
  Time to nadir, Hemoglobin | 49.5 (27.53)
  Time to nadir, Platelet count | 35.5 (6.94)
  Time to nadir, WBC count | 52.7 (16.28)

11. Secondary Outcome: Number of Participants Needing Supportive Care at Week 7 and Week 13
Description: During the administration of unlabeled Anti-B1 antibody and Iodine-131 Anti-B1 antibody, emergency support for anaphylaxis, including epinephrine, diphenhydramine, hydrocortisone, a laryngoscope, and an endotracheal tube, was readily available. The use of steroids were discouraged unless other measures were ineffective.
Time Frame: Week 7 and Week 13
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
participants
  Week 7, any supportive care | 3
  Week 13, any supportive care | 3

12. Secondary Outcome: Number of Participants Converting to Human Anti-Murine (Mouse) Antibody (HAMA) Positivity at Any Follow-up Visit From HAMA Negativity at Baseline
Description: The number of participants who developed human anti-murine (mouse) anibodies (HAMA) after treatment was measured.
Time Frame: Baseline; any follow-up visit (up to 72 months)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
participants
  Positive | 1
  Negative | 14

13. Secondary Outcome: Overall Survival
Description: Overall survival (time to death) is defined from the start of treatment to the date of death from any cause.
Time Frame: From Baseline until Week 25 and follow-up (up to 130 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST/Iodine I-131 TST
Number analyzed (Participants) | 15
months | NA [NA to NA] — Median overall survival could not be estimated by the Kaplan-Meier method because the median was not reached.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the treatment period (up to 130 months).
Description: An on-therapy AE or SAE is defined as an AE with an onset on or after the start date of study medication, but not later than one day after the last date of study medication. SAEs and AEs were collected in members of the ITT Population, comprised of all participants who received study drug.
Arm/Group | TST/Iodine I-131 TST
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST/Iodine I-131 TST (N=15)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Central nervous system lesion (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST/Iodine I-131 TST (N=15)
Fatigue (General disorders) | 11
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Local swelling (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
ANC (calc) < 1,000 cells/mm3 (Investigations) | 7
WBC < 2,000 cells/mm3 (Investigations) | 6
Platelets <50,000 cells/mm3 (Investigations) | 4
Hemoglobin <8.0 gm/dL (Investigations) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 2
Burning sensation (Nervous system disorders) | 1
Central nervous system lesion (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Candidiasis (Infections and infestations) | 1
Fungal infection (Congenital, familial and genetic disorders) | 1
Herpes zoster (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Blood pressure decreased (Investigations) | 1
Blood urine present (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ear pain (Ear and labyrinth disorders) | 1
Lacrimation increased (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Affect lability (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.